CLINICAL TRIAL: NCT06927700
Title: Effects of FDA Authorized Smokeless Tobacco Claims Among US Adults Who Smoke Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olivia A. Wackowski, PhD, MPH, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2024000097; R21CA289541 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Product Beliefs and Use
Keywords: smokeless tobacco; tobacco advertising; modified risk claims; snus; moist snuff
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (General Snus-Control Ads) (Other): Participants in this group will view 4 ads for the brand General Snus that do not include a modified risk claim.
  Interventions: Behavioral: Modified Risk Claim Type - None; Behavioral: Product Brand - General Snus
- Group 2 (General Snus-Multiple Disease Ads) (Experimental): Participants in this group will view 4 ads for the brand General Snus that include a modified risk claim about the lower risk of multiple diseases.
  Interventions: Behavioral: Product Brand - General Snus; Behavioral: Modified Risk Claim Type - Multiple Diseases
- Group 3 (General Snus- Lung Ads) (Experimental): Participants in this group will view 4 ads for the brand General Snus that include a modified risk claim about the lower risk of lung cancer only.
  Interventions: Behavioral: Product Brand - General Snus; Behavioral: Modified Risk Claim Type - Lung Cancer
- Group 4 (Copenhagen-Control Ads) (Experimental): Participants in this group will view 4 ads for the brand Copenhagen that do not include a modified risk claim.
  Interventions: Behavioral: Modified Risk Claim Type - None; Behavioral: Product Brand - Copenhagen
- Group 5 (Copenhagen-Multiple Disease Ads) (Experimental): Participants in this group will view 4 ads for the brand Copenhagen that include a modified risk claim about the lower risk of multiple diseases.
  Interventions: Behavioral: Product Brand - Copenhagen; Behavioral: Modified Risk Claim Type - Multiple Diseases
- Group 6 (Copenhagen- Lung Ads) (Experimental): Participants in this group will view 4 ads for the brand Copenhagen that include a modified risk claim about the lower risk of lung cancer only.
  Interventions: Behavioral: Product Brand - Copenhagen; Behavioral: Modified Risk Claim Type - Lung Cancer

INTERVENTIONS:
Behavioral: Modified Risk Claim Type - None — Participants will view smokeless tobacco ads with no modified risk claim (control)
  Arms: Group 1 (General Snus-Control Ads); Group 4 (Copenhagen-Control Ads)
Behavioral: Product Brand - General Snus — Participants will views ads for the smokeless tobacco brand General Snus
  Arms: Group 1 (General Snus-Control Ads); Group 2 (General Snus-Multiple Disease Ads); Group 3 (General Snus- Lung Ads)
Behavioral: Product Brand - Copenhagen — Participants will views ads for the smokeless tobacco brand Copenhagen
  Arms: Group 4 (Copenhagen-Control Ads); Group 5 (Copenhagen-Multiple Disease Ads); Group 6 (Copenhagen- Lung Ads)
Behavioral: Modified Risk Claim Type - Multiple Diseases — Participants will view smokeless tobacco ads with a claim about lower risks for multiple diseases
  Arms: Group 2 (General Snus-Multiple Disease Ads); Group 5 (Copenhagen-Multiple Disease Ads)
Behavioral: Modified Risk Claim Type - Lung Cancer — Participants will either view smokeless tobacco ads with a modified risk claim about lower risks for lung cancer only
  Arms: Group 3 (General Snus- Lung Ads); Group 6 (Copenhagen- Lung Ads)

SUMMARY:
This study will be an online survey experiment conducted with adults who smoke cigarettes (ages 21+) to examine their reactions to modified risk advertising claims authorized by the Food & Drug Administration (FDA) for two smokeless tobacco brands (General Snus and Copenhagen), which describe the lower risks of these products compared to cigarette smoking. The study will compare effects of ads with different two different claim types (i.e. claims about reduced lung cancer risk and claims about reduced risks for multiple disease) versus ads with no reduced-risk claims, and examine effects on message and product perceptions, and interest in using the smokeless tobacco products. This study will also examine how smokers' reactions/interest may vary based on the product brand, and asses prior awareness/exposure to the authorized claims.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 21 and over) who are current established cigarettes smokers (i.e., smoked 100 cigarettes in their lifetime and now smoke every day or somedays), based in the US, members of Ipsos' KnowledgePanel, and have chosen to complete their research panel surveys in English

Exclusion Criteria:

* Panel participants who do not meet the criteria outlined above will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Product Relative Harm/Risk Perceptions | Assessed in survey measures completed immediately after viewing the study stimuli
  Multi-item assessment of perceived harm/risks from using the smokeless tobacco products viewed as compared smoking cigarettes
Product Use Intentions | Assessed in survey measures completed immediately after viewing the study stimuli
  Multi-item assessment of intentions to use the viewed smokeless tobacco products, including interest in trying the product, switching to the product, and likelihood of buying the product

SECONDARY OUTCOMES:
Message Recall | Assessed in survey measures completed immediately after viewing the study stimuli
  Participants will be asked if they recall (yes/no) if the ads made any risk comparisons with cigarettes, and, if yes, to describe these in an open-ended measure, followed by an aided recall item (with correct and incorrect claim options).
Add and message perceptions | Assessed in survey measures completed immediately after viewing the study stimuli
  Multi-item assessments to rate the ad stimuli and modified risk claim on perceptions such as believability, credibility, importance, understandability, novelty, and perceived impact on interest in learning more about the products and wanting to use the products
Switching comprehension | Assessed in survey measures completed immediately after viewing the study stimuli
  An item to assess participants' understanding of the need to completely switch to the smokeless tobacco product in order to reduce risks.
Main cause of smoking harms | Assessed in survey measures completed immediately after viewing the study stimuli
  An item to explore understanding of the main source of harm from smoking cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia A Wackowski, PhD, MPH, Principal Investigator — Rutgers University
Locations (1):
- Rutgers Institute for Nicotine & Tobacco Studies, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The study ad stimuli, survey instrument, codebook, and de-identified dataset will be deposited to a data repository - we anticipate this will be the National Addiction and HIV Data Archive Program (NAHDAP), currently managed by ICPSR at the University of Michigan.
Supporting Information: Analytic Code
Time Frame: The scientific community will be able to access the data at the end of the award period. All publications using the data will also reference the data location in NAHDAP/ICSPR using DOIs. ICPSR engages in long-term preservation of the research data upon receipt of a signed deposit form, including migration to new formats, platforms, and storage media as required. ICPSR has a commitment to designate a successor repository in the unlikely event that such a need arises.
Access Criteria: To request access, interested researchers will use the standard processes at NAHDAP/ICSPR for requesting data.

REFERENCES:
- See also: Information about FDA's authorization of modified risk order for Copenhagen snuff — https://www.fda.gov/tobacco-products/advertising-and-promotion/us-smokeless-tobacco-company-modified-risk-tobacco-product-mrtp-application
- See also: Information about FDA's authorization of modified risk order for General Snus products — https://www.fda.gov/tobacco-products/fda-renews-authorization-8-general-snus-products-be-marketed-reduced-risk-claim

DOCUMENTS (1):
  • Informed Consent Form (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT06927700/ICF_000.pdf